CLINICAL TRIAL: NCT05813678
Title: A Multi-Center, Observational Study to Evaluate the Long-Term Safety of Subcutaneous Injections of Palynziq® (Pegvaliase) in Subjects With Phenylketonuria
Brief Title: A Long-term, Post-marketing Safety Study of Palynziq in Patients With PKU (PALace)
Acronym: PALace
Status: Recruiting | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 165-501; EUPAS34992 (Registry Identifier: European Network of Centres for Pharmacoepidemiology and Pharmacovigilance)
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Phenylketonuria (PKU)
Keywords: Observational; Safety Study; Pegvaliase; Palynziq; PKU; Phenylketonuria; Phase 4
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pegvaliase — This is an uncontrolled, single-cohort, Phase 4 observational study not falling under the definition of an Applicable Clinical Trial (ACT) (i.e., non-interventional).

SUMMARY:
This is a 10-year multi-center, global, observational study to further characterize the safety profile of pegvaliase, including hypersensitivity reactions, long-term safety and tolerability, and the effectiveness of the additional risk minimization measures (aRMMs) (European Union (EU) only) in subjects receiving pegvaliase for the treatment of PKU. Subjects for whom a clinical decision has been made that they will receive pegvaliase to treat their PKU within 30 days following the date of enrollment (incident-users) or have previously started treatment with pegvaliase at the date of enrollment (prevalent-users) are eligible for participation in this study.

DETAILED DESCRIPTION:
This is a 10-year multi-center, global, observational study to further characterize the safety profile of pegvaliase, including hypersensitivity reactions, long-term safety and tolerability, and the effectiveness of the aRMMs (EU only) in subjects receiving pegvaliase for the treatment of PKU. Subjects for whom a clinical decision has been made that they will receive pegvaliase to treat their PKU within 30 days following the date of enrollment (incident-users) or have previously started treatment with pegvaliase at the date of enrollment (prevalent-users) are eligible for participation in this study. Once the subject has been enrolled, the investigator (ie, subject's primary physician) will be asked to provide information about the subject's medical history, treatment(s) received to manage their blood Phe levels, treatment with pegvaliase, and concomitant medication use. The investigator will also be asked to provide evaluation of the following safety concerns: Acute systemic hypersensitivity reaction, Anaphylaxis, Angioedema, Serum sickness, Severe hypersensitivity reaction, Severe or Persistent arthralgia, Severe injection site reaction, Hypophenylalaninemia and other protocol-defined safety events, following the initiation of pegvaliase therapy. There are no protocol-mandated visits or procedures associated with this study. Enrolled subjects should be followed per routine clinical practice at the institution based upon their diagnosis, with clinical outcomes assessed at regular intervals (typically every month during the induction and titration phases of pegvaliase treatment and every 6 months once the maintenance phase is reached). No experimental treatment or assessments are planned as part of this observational study. An Independent Adjudication Committee (IAC) will periodically review protocol-defined safety events, including Acute systemic hypersensitivity reaction and Serum sickness.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of PKU per local standard of care
* Currently receiving or planned to receive pegvaliase treatment within 30 days after the date of enrollment, including subjects who previously received pegvaliase as part of the clinical development program and have completed study participation.
* Subject (or legally authorized representative) is willing and able to provide written informed consent after the nature of the study has been explained and prior to any data collection.

Exclusion Criteria:

* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with any aspect of the study.
* Currently participating in an interventional study of any investigational product, device, or procedure
* Previously enrolled in this study (eg, subjects who have been withdrawn from the study and wish to participate again at a later date)
* German subjects <16 years if age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects with PKU followed at participating centers, currently receiving or planning to receive pegvaliase treatment.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2033-11-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
To quantify and characterize the risk of protocol-defined safety events in incident-users receiving pegvaliase for the treatment of PKU in a real¬ world setting. | A maximum of 10 years treatment duration.
  Analyses on incident-users are considered primary. The primary analysis is the incidence rate of:
  Acute systemic hypersensitivity reaction
  Anaphylaxis
  Angioedema
  Serum sickness
  Severe hypersensitivity reaction
  Severe or Persistent (≥ 6 months) or arthralgiaSevere injection site reactionHypophenylalaninemia.

SECONDARY OUTCOMES:
To quantify and characterize the risk of protocol-defined safety events in subjects receiving pegvaliase for the treatment of PKU in a real-world setting. | A maximum of 10 years treatment follow up duration.
  Secondary analyses under safety events will include:
  The incidence rate of:
  * End-organ damage associated with immune-complex formation, or PEG accumulation.
  * SAEs• Severe ADRs
  * ADRs leading to treatment interruption or discontinuation and/or study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (16):
- United States (8):
  - University of Colorado, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (4):
  - Hospital Carl-Thiem-Klinikum Cottbus, Cottbus
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Münster (UKM)-Pädiatrische Universitätsklinik Münster, Münster
  - Universität Ulm, Ulm
- Italy (4):
  - Policlinico Sant'orsola Malpighi, Bologna
  - University Hospital Careggi, Florence
  - Ospedale San Paolo, Milan
  - Azienda Ospedaliera Universitaria "Federico II" Dipartimento di Pediatria, Naples